CLINICAL TRIAL: NCT02590510
Title: Different Dose of Methotrexate for the Treatment of Meningeal Carcinomatosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hui Bu (Other)
Responsible Party: Sponsor-Investigator, Hui Bu, Study Principal Investigator, Hebei Medical University
Organization: Hebei Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BH 001
Record Dates: First submitted 2015-10-26; First posted 2015-10-29 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Meningeal Carcinomatosis
Keywords: Intrathecal chemotherapy
MeSH Terms: conditions — Meningeal Carcinomatosis | interventions — Methotrexate

ARMS (2):
- The small dose of group (Experimental): The dose of methotrexate is 10 mg
  Interventions: Drug: methotrexate
- The high dose of group (Active Comparator): The dose of methotrexate is 15 mg
  Interventions: Drug: methotrexate

INTERVENTIONS:
Drug: methotrexate — The quantity of methotrexate is different in the two groups.
  Other Names: Intrathecal chemotherapy

SUMMARY:
The main purpose of this study is to compare the effect of 10 mg and 15 mg methotrexate in the treatment of meningeal carcinomatosis.

ELIGIBILITY:
Inclusion Criteria:

* age 14 or more
* a history of solid tumor
* a new clinical neurological signs and symptoms
* a typical CT(Computerized Tomography,CT) or MRI(Magnetic Resonance Imaging,MRI) imaging findings
* tumor cells in cerebrospinal fluid

Exclusion Criteria:

* KPS score <60
* the tumor patients with organ failure
* bacteria, fungi or viral meningitis

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
overall survival | one year

SECONDARY OUTCOMES:
The incidence of adverse reactions | one year
  In accordance with the standard of CTCAE, an assessment will be assessed every month
KPS score | one year
  In accordance with the standard of KPS(Karnofsky Performance Status,KPS) score, an assessment will be assessed every month

CONTACTS AND LOCATIONS:
Overall Officials: Hui, Principal Investigator — The Second Hospital of Hebei Medical University